CLINICAL TRIAL: NCT01329146
Title: Pulse Pressure Variations as Index of Preload Dependency During Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-A00302-53; PROM 2008/0812 (Other: Sponsor)
Record Dates: First submitted 2011-04-04; First posted 2011-04-05 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Fluid Response
Keywords: pulse pressure variation; preload dependency; one-lung ventilation; thoracic surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: calculation of the pulse pressure variation (PPV) has repeatedly been shown to be a reliable predictor of fluid responsiveness in mechanically ventilated patients. But PPV measurement has not been yet validated in thoracic surgery during one-lung ventilation. The modifications of intrathoracic pressure induced by one-lung ventilation may altered the capabilities of PPV to predict fluid responsiveness.This study was designed to assess the ability of PPV predict fluid responsiveness during one-lung ventilation in thoracic surgery.

Methods: a prospective observational study. Thirty five patients undergoing a pulmonary resection (lobectomy or pneumonectomy) will be included to achieve around one hundred fluid challenges with a 250 milliliters colloid solution in response to hemodynamic instability.Hemodynamic instability is defined as a decrease by 20 % of artery pressure from baseline and/or an increase by 20% heart rate from baseline. Fluid responsiveness is defined as an increase in stroke volume index (SVI)>10% (measured with oesophageal doppler). PPV will be calculated from recorded artery pressure curve (PPVref) before and after each fluid challenge. An automated measurement of PPV proposed by the monitor Intelview (Philips) will be recorded simultaneously before and after each fluid challenge.

Statistical analysis: receiver operating characteristic curve will be used to assess the PPV capability to predict fluid responsiveness. Correlation analysis will be achieved using a Pearson test or Spearman's rho test when necessary. Continuous data will compared using a Student t test or a Mann-Whitney test when necessary.

DETAILED DESCRIPTION:
* pulse pressure variation
* preload dependency
* one-lung ventilation
* thoracic surgery

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing a thoracic surgery (lobectomy, bilobectomy or pneumonectomy).
* All patients requiring a hemodynamic monitoring (artery catheter, oesophageal doppler).

Exclusion Criteria:

* Arrythmia.
* Pregnant patient.
* Patients less than 18 years old.
* oesophageal or gastric pathologies precluding the use of oesophageal doppler.
* pathologies precluding the use of artery catheter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing a thoracic surgery (lobectomy or pneumonectomy)and requiring hemodynamic monitoring (artery catheter, oesophageal doppler)in the thoracic surgery unit of the university hospital of Lille.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel ROBIN, MD PhD, Principal Investigator — Reanimation Department, University Hospital of Lille
Locations (1):
- Thoracic surgery department, University Hospital of Lille, Lille, France

IPD SHARING:
Plan to Share IPD: Undecided